CLINICAL TRIAL: NCT06188052
Title: Efficacy of Topical Versus Intravenous Tranexamic Acid in Controlling Blood Loss in Patients Undergoing:Total Laryngectomy With Neck Dissection. A Randomized Control Study.
Brief Title: Efficacy of Topical Versus Intravenous Tranexamic Acid in Controlling Blood Loss
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Dina Mahmoud Mohamed, Lecturer of Anesthesia and Surgical ICU and pain management, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-97-2023
Record Dates: First submitted 2023-09-19; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: To Calculate Total Blood Loss Immediately Postoperative
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: All procedures will be performed by the same team, all of whom will be blind to the group assignment (except for the resident who will prepare the drug formula whether intravenous or the topical irrigation and will be responsible for randomization and drug masking using closed envelope randomization)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A), tranexamic acid IV (Active Comparator): tranexamic acid will be given 1 hr preoperatively as 1mg/kg intravenously
  Interventions: Drug: Tranexamic acid
- Group (B), topical tranexamic acid (Active Comparator): topical tranexamic acid will be given as an irrigation by 40 ml of tranexamic acid 2mg/kg dissolved in 200ml to the surgical site every 1 hour for the first 5 hours .
  Interventions: Drug: Tranexamic acid
- Group (C), control group. (Placebo Comparator): Saline will be given intravenously instead of tranexamic acid And irrigation with Saline instead of tranexamic acid
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — Comparing the 3 groups regarding intraoperative bleeding, hemoglobin level pre and postoperative and the need of blood transfusion

SUMMARY:
Total laryngectomy with bilateral block neck dissection is considered one of the major head and neck surgeries. Intraoperative bleeding is considered a risk factor for this operation specially that the population of this operation are elder with multiple comorbidities. Intravenous administration of tranexamic acid reduces bleeding during surgery.We design this study aiming to prove the role of topical tranexamic acid in controlling the intraoperative bleeding in patients undergoing total laryngectomy operation avoiding the risk of intravenous administration.

DETAILED DESCRIPTION:
45 patients undergoing total laryngectomy operation will be enrolled in this study. The patients will be divided into 3 equal groups, 15 patients in each group. Group (A), tranexamic acid will be given 1 hr preoperatively. Group (B), topical tranexamic acid will be given as an irrigation to the surgical site. Group (C), control group.One hour preoperatively, a wide bore cannula will be inserted to all patients. Tranexamic acid 1mg/kg will be given intravenously to patients in group (A). Normal saline will be given to Group (B) and group (C) .On arrival to the operating room, a pulse oximetry, continuous electrocardiogram (ECG), and non-invasive blood pressure measurement device will be connected to the patient. Pre-medications will be given; metoclopramide (10mg) and dexamethasone (8mg) preoperatively. Induction will be done by sevoflurane, propofol 1mg/ kg, succinyl choline 0.5mg/kg. After intubation, fentanyl 2mic/kg and atracurium 0.5mg/kg will be given , followed by 0.8 mg/kg Morphine sulphate . Anesthesia will be maintained by isoflurane 1.5% and atracurium 0.1mg/kg/ 30min. After flap elevation ( using local infiltraton of epinephrine 1/100000), the surgical site will be irrigated by 40 ml of tranexamic acid 2mg/kg dissolved in 200ml normal saline every 1 hour for the first 5 hours in group (B), and by normal saline in group (A) and group (C).

ELIGIBILITY:
Inclusion criteria:

- Patients of either sex, aged between 18-70 years old, ASA physical status I, II undergoing total laryngectomy

Exclusion Criteria:

* Patients with coagulopathy, a history of thromboembolism or a history of tranexamic acid allergy or complication will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
To calculate total blood loss immediately postoperative and compare it in 3 groups To calculate total blood loss and compare 3 groups | Intraoperative
  Intraoperative bleeding will be assessed and blood loss will be measured in ml ( amount of blood in canister and sponges)

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Mohamed, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University hospitals, Cairo, Egypt